CLINICAL TRIAL: NCT02094716
Title: A Multicenter, Randomized, Double-Blind, Parallel Group Comparison Study of the Safety and Efficacy of Permethrin Foam, 5% Versus Permethrin Foam, 4% Versus Vehicle in Subjects With Sarcoptes Scabiei
Brief Title: A Dose Ranging Vehicle Controlled Study to Determine the Safety and Efficacy of Permethrin Foam, 5% and Permethrin Foam, 4% for the Treatment of Scabies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: DPT Laboratories, Ltd. (Industry); Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 185-7851-201
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Scabies
Keywords: Sarcoptes; Scabiei; Scabies; ectoparasite; parasite; infestation; Renaissance
MeSH Terms: conditions — Scabies; Parasitic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Permethrin Foam 4%/ Permethrin Foam 4% (Experimental): First treatment with Permethrin Foam 4% with potential to re-treat with Permethrin Foam 4%, if necessary.
  Interventions: Drug: Permethrin Foam 4%
- Permethrin Foam 5%/ Permethrin Foam 5% (Experimental): First treatment with Permethrin Foam 5% with potential to re-treat with Permethrin Foam 5%, if necessary.
  Interventions: Drug: Permethrin Foam 5%
- Vehicle Foam / Permethrin Foam 4% (Placebo Comparator): First treatment with Vehicle with potential to re-treat with Permethrin Foam 4%, if necessary.
  Interventions: Drug: Permethrin Foam 4%; Drug: Vehicle Foam
- Vehicle / Permethrin Foam 5% (Placebo Comparator): First treatment with Vehicle with potential to re-treat with Permethrin Foam 5%, if necessary.
  Interventions: Drug: Permethrin Foam 5%; Drug: Vehicle Foam

INTERVENTIONS:
Drug: Permethrin Foam 4% — Topical application, whole-body treatment
  Other Names: PF-045
  Arms: Permethrin Foam 4%/ Permethrin Foam 4%; Vehicle Foam / Permethrin Foam 4%
Drug: Permethrin Foam 5% — Topical application, whole-body treatment
  Other Names: PF-055
  Arms: Permethrin Foam 5%/ Permethrin Foam 5%; Vehicle / Permethrin Foam 5%
Drug: Vehicle Foam — Topical application, whole-body treatment
  Other Names: Vehicle
  Arms: Vehicle / Permethrin Foam 5%; Vehicle Foam / Permethrin Foam 4%

SUMMARY:
To determine and compare the safety and efficacy of permethrin foam 4% and permethrin foam 5% with that of vehicle in subjects with scabies.

DETAILED DESCRIPTION:
It is anticipated that a majority of subjects will require and receive a single treatment; however, those subjects not showing improvement at the follow-up visit 2 weeks after initial treatment will be treated a second time. Those subjects originally assigned to vehicle for the first treatment will receive a "re-treatment" with one of the active doses.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of active scabies infection.
* Subject is in good general health with normal appearing skin in noninfested areas.
* Females must be post-menopausal, surgically sterile or use an effective method of birth control with a negative pregnancy test (10 years of age and older) at study start.

Exclusion Criteria:

* Subject is pregnant, lactating, or is planning to become pregnant during the study.
* Subject has used any ectoparasiticide within the three weeks prior to study start.
* Subject has signs of systemic infection or is receiving systemic therapy for an infectious disease.
* Subject has severe cutaneous bacterial or fungal infections requiring therapy or heavily crusted lesions consistent with Norwegian scabies.
* Subject is currently enrolled in an investigational drug or device study or has used an investigational drug or device within 30 days prior to study start.
* Subject whose close personal contacts will not comply with standard of care for fomite management.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - Clinical Research Site, Fremont, California
  - Clinical Research Site, Los Angeles, California
  - Clinical Research Site, Hialeah, Florida
  - Clinical Research Site, New York, New York
  - Clinical Research Site, Philadelphia, Pennsylvania
- Dominican Republic (2):
  - Clinical Research Site, San Cristóbal
  - Clinical Research Site, Santo Domingo
- Clinical Research Site, San Pedro Sula, Honduras
- Clinical Research Site, Ponce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- Permethrin Foam 4%/ Permethrin Foam 4%: First treatment with Permethrin Foam 4% with potential to re-treat with Permethrin Foam 4%, if necessary.
  Topical application, whole-body treatment
- Permethrin Foam 5%/ Permethrin Foam 5%: First treatment with Permethrin Foam 5% with potential to re-treat with Permethrin Foam 5%, if necessary.
  Topical application, whole-body treatment
- Vehicle Foam: First treatment with Vehicle with potential to re-treat with Permethrin Foam, if necessary.
  Topical application, whole-body treatment
Period: Overall Study
Arm/Group | Permethrin Foam 4%/ Permethrin Foam 4% | Permethrin Foam 5%/ Permethrin Foam 5% | Vehicle Foam
Started | 43 | 43 | 44
Received Second Dose at Day 14 (Of 44 subjects who had a first dose of vehicle, 8 received a second treatment with 4% and 9 with 5%.) | 15 | 10 | 17
Completed | 41 | 36 | 40
Not Completed | 2 | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Permethrin Foam 4%/ Permethrin Foam 4% | Permethrin Foam 5%/ Permethrin Foam 5% | Vehicle Foam | Total
Number analyzed (Participants) | 43 | 43 | 44 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (20.8) | 23.4 (18.4) | 26.1 (20.4) | 25.9 (19.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 19 | 61
  Male | 19 | 25 | 25 | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Received a Single Treatment of the Assigned Test Article That Were Designated as "Treatment Success"
Description: The primary efficacy variable is "treatment success". In protocol v2.0, "treatment success" was defined as an Investigator's Global Assessment (IGA) score of 0 (clear) or 1 (almost clear). In protocol v3.0, "treatment success" was defined as an "eradication of infestation": a) no burrows, b) a reduction in the Signs/Symptoms, and c) no evidence of a live mite on microscopy.
Time Frame: Day 28
Population: Intent to Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Permethrin Foam 4%/ Permethrin Foam 4% | Permethrin Foam 5%/ Permethrin Foam 5% | Vehicle Foam
Number analyzed (Participants) | 43 | 43 | 44
Participants | 23 | 26 | 22
Statistical Analysis 1: Comparison: Permethrin Foam 4%/ Permethrin Foam 4% vs Permethrin Foam 5%/ Permethrin Foam 5% vs Vehicle Foam; Test type: Superiority; p = 0.6084, Chi-squared

2. Secondary Outcome: Change in Disease-related Signs and Symptoms for Those Subjects Provided With Re-treatment at Day 14 Who Show Improvement in Their Investigator's Global Assessment (IGA) Score at Day 28
Description: The change in the total score of signs and symptoms related to the condition in each treatment group at Days 14 and 28, as well as at Day 42 for those subjects provided with re-treatment at Day 14 who show improvement in their IGA score at Day 28.
  Scale details: The overall average presence of the individual signs and symptoms of scabies was evaluated over the entire body. Erythema, papules, pustules, crusting, scaling, excoriations, and pruritus were assessed as follows for each sign and symptom: None=0, Trace=1, Mild=2, Moderate=3, Severe=4. From these assessments, the total score of the Signs and Symptoms (from 0 to 28, higher scores mean a worse outcome) was calculated as the sum of the individual signs and symptoms scores at Baseline and Days 2, 14, 28, and 42 (if applicable).The change from baseline in the total score can range from -28 as the best reduction possible (better outcome) to +28 as the worst increase possible (worse outcome) in signs and symptoms.
Time Frame: Baseline, Day 14, 28, and 42
Population: Missing data not included
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Permethrin Foam 4%; Permethrin Foam 4%: First treatment with Permethrin Foam 4% with re-treatment with Permethrin Foam 4% at Day 14 who were also improving at Day 28.
  Topical application, whole-body treatment
- Permethrin Foam 5%; Permethrin Foam 5%: First treatment with Permethrin Foam 5% with re-treatment with Permethrin Foam 5% at Day 14 who were also improving at Day 28.
  Topical application, whole-body treatment
- Vehicle; Permethrin Foam 4%: First treatment with Vehicle Foam with second treatment with Permethrin Foam 4% at Day 14 who were also improving at Day 28
  Topical application, whole body treatment
- Vehicle Foam; Permethrin Foam 5%: First treatment with Vehicle with second treatment of Permethrin Foam 5% at Day 14 who were also improving at Day 28.
  Topical application, whole-body treatment
Arm/Group | Permethrin Foam 4%; Permethrin Foam 4% | Permethrin Foam 5%; Permethrin Foam 5% | Vehicle; Permethrin Foam 4% | Vehicle Foam; Permethrin Foam 5%
Number analyzed (Participants) | 10 | 7 | 7 | 7
score on a scale
  Day 14 Change from Baseline | -1.1 (2.7) | 0.6 (2.0) | -0.1 (2.5) | 0.6 (3.5)
  Day 28 Change from Prior Visit (Day 14): number analyzed (Participants) | 10 | 6 | 7 | 7
  Day 28 Change from Prior Visit (Day 14) | -11.2 (4.5) | -9.0 (5.9) | -11.4 (6.7) | -9.7 (7.7)
  Day 42 Change from Prior Visit (Day 28): number analyzed (Participants) | 10 | 4 | 5 | 5
  Day 42 Change from Prior Visit (Day 28) | -0.5 (4.0) | -2.5 (2.9) | -2.4 (2.4) | -3.4 (6.6)

3. Secondary Outcome: Number of Re-treated Subjects Designated as "Treatment Success"
Description: Each subject was designated as "re-treatment success" at Day 42 based upon the criteria in the protocol to which he/she was enrolled. In protocol v2.0, "treatment success" was defined as an Investigator's Global Assessment (IGA) score of 0 (clear) or 1 (almost clear). In protocol v3.0, "treatment success" was defined as an "eradication of infestation": a) no burrows, b) a reduction in the Signs/Symptoms, and c) no evidence of a live mite on microscopy.
Time Frame: Day 42
Population: ITT subjects who did not improve at Day 14 and received a second treatment at Day 14
Measure: Count of Participants; unit: Participants
Groups:
- Permethrin Foam 4%; Permethrin Foam 4%: First treatment with Permethrin Foam 4% with potential to re-treat with Permethrin Foam 4%, if necessary.
  Topical application, whole-body treatment
- Permethrin Foam 5%; Permethrin Foam 5%: First treatment with Permethrin Foam 5% with potential to re-treat with Permethrin Foam 5%, if necessary.
  Topical application, whole-body treatment
- Vehicle Foam; Permethrin Foam 4%: First treatment with Vehicle with potential to re-treat with Permethrin Foam 4%, if necessary.
  Topical application, whole-body treatment
- Vehicle; Permethrin Foam 5%: First treatment with Vehicle with potential to re-treat with Permethrin Foam 5%, if necessary.
  Topical application, whole-body treatment
Arm/Group | Permethrin Foam 4%; Permethrin Foam 4% | Permethrin Foam 5%; Permethrin Foam 5% | Vehicle Foam; Permethrin Foam 4% | Vehicle; Permethrin Foam 5%
Number analyzed (Participants) | 10 | 7 | 7 | 7
Participants | 8 | 4 | 5 | 4
Statistical Analysis 1: Comparison: Permethrin Foam 4%; Permethrin Foam 4% vs Permethrin Foam 5%; Permethrin Foam 5% vs Vehicle Foam; Permethrin Foam 4% vs Vehicle; Permethrin Foam 5%; Test type: Superiority; p = 0.6937, Chi-squared

4. Secondary Outcome: Number of Subjects Designated as "Treatment Success" Following One Treatment With an Active Dose
Description: The proportion of subjects designated as "treatment success" following one treatment versus two treatments.
  In protocol v2.0, "treatment success" was defined as an Investigator's Global Assessment (IGA) score of 0 (clear) or 1 (almost clear). In protocol v3.0, "treatment success" was defined as an "eradication of infestation": a) no burrows, b) a reduction in the Signs/Symptoms, and c) no evidence of a live mite on microscopy.
  Subjects originally assigned to vehicle treatment and re-treated on Day 14 with an active dose will be included with the single treatment group for this analysis.
  Subjects who did not improve at Day 14 were counted as failures at Day 28. Subjects who improved at Day 14 and received a second treatment in error were counted as failures at Day 28.
Time Frame: Day 28 and Day 42
Measure: Count of Participants; unit: Participants
Groups:
- Permethrin Foam 4% Two Active Treatments: First treatment with Permethrin Foam 4%, second treatment with Permethrin Foam 4%.
  Topical application, whole-body treatment
- Permethrin Foam 5% Two Active Treatments: First treatment with Permethrin Foam 5%, second treatment with Permethrin Foam 5%.
  Topical application, whole-body treatment
- Permethrin Foam 4% Single Active Treatment: If the subject was improved at Day 14 and only received one treatment (Permethrin Foam, 4%), or if the subject received Vehicle Foam at Baseline, was not improved at Day 14, and received a single active (Permethrin Foam, 4%) treatment at Day 14.
  Topical application, whole-body treatment
- Permethrin Foam 5% Single Active Treatment: If the subject was improved at Day 14 and only received one treatment (Permethrin Foam, 5%), or if the subject received Vehicle Foam at Baseline, was not improved at Day 14, and received a single active (Permethrin Foam, 5%) treatment at Day 14.
  Topical application, whole-body treatment
Arm/Group | Permethrin Foam 4% Two Active Treatments | Permethrin Foam 5% Two Active Treatments | Permethrin Foam 4% Single Active Treatment | Permethrin Foam 5% Single Active Treatment
Number analyzed (Participants) | 15 | 10 | 36 | 42
Participants | 8 | 4 | 28 | 30
Statistical Analysis 1: Comparison: Permethrin Foam 4% Two Active Treatments vs Permethrin Foam 4% Single Active Treatment; Test type: Superiority; p = 0.1010, Fisher Exact
Statistical Analysis 2: Comparison: Permethrin Foam 5% Two Active Treatments vs Permethrin Foam 5% Single Active Treatment; Test type: Superiority; p = 0.0764, Fisher Exact

ADVERSE EVENTS:
Description: Subjects randomized to Vehicle/Permethrin Foam, 5% or Vehicle/Permethrin Foam, 4% who received a second treatment are counted in the Permethrin Foam, 5% or Permethrin Foam, 4% and Vehicle treatment groups. For subjects randomized to Vehicle Foam on Day 1 who were re-treated at Day 14 (Visit 3), Adverse Events (AEs) were assigned to Vehicle Foam group if the event occurred before Day 14 (Visit 3) or to the active treatment group if the event took place after Day 14 (Visit 3).
Groups:
- Permethrin Foam 4%: Treatment with Permethrin Foam 4%.
  Topical application, whole-body treatment
- Permethrin Foam 5%: Treatment with Permethrin Foam 5%.
  Topical application, whole-body treatment
- Vehicle Foam: Treatment with Vehicle Foam.
  Topical application, whole-body treatment
Arm/Group | Permethrin Foam 4% | Permethrin Foam 5% | Vehicle Foam
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/52 | 0/44
Other Adverse Events (participants affected / at risk) | 0/51 | 0/52 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event said right to publish is exercised, the Investigator shall submit to Sponsor for review 60 days prior to any publication. In the event that Sponsor desires to take patent action, Investigator agrees to delay the publication an additional 60 days. Sponsor shall have the right to review and comment upon such publication. Notwithstanding the foregoing, no paper that incorporates Sponsor Confidential Information shall be submitted for publication without Sponsor's prior written consent.